CLINICAL TRIAL: NCT03406312
Title: European Dumping Study: Validation of a Diagnostic Tool for Postprandial Hypoglycaemia in Patients After Roux en Y Gastric Bypass Surgery
Brief Title: Validation of a Diagnostic Tool for Postprandial Hypoglycaemia in Patients After Roux en Y Gastric Bypass Surgery
Acronym: EDS
Status: Completed | Type: Observational
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: B670201731703
Record Dates: First submitted 2018-01-12; First posted 2018-01-23 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Post Prandial Hypoglycemia
Keywords: Roux en Y Gastric Bypass Surgery, Hypoglycemia, Postprandial
MeSH Terms: conditions — Hypoglycemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Gastric Bypass Surgery population: liquid mixed meal tolerance test, solid mixed meal tolerance test, continuous glucose monitoring
  Interventions: Diagnostic Test: Post Prandial Hypoglycemia test
- Control population: liquid mixed meal tolerance test, solid mixed meal tolerance test, continuous glucose monitoring
  Interventions: Diagnostic Test: Post Prandial Hypoglycemia test

INTERVENTIONS:
Diagnostic Test: Post Prandial Hypoglycemia test — three test assessing hypoglycemia will be used: liquid mixed meal tolerance test, solid mixed meal tolerances test, continuous glucose monitoring

SUMMARY:
Roux-en-Y gastric bypass (RYGB) leads to weight reduction but has also some unwanted side effects. A part of this population will develop postprandial reactive hypoglycemia (PPRH). At this moment no validated diagnostic tool exists for PPRH. The aim of this study is to prove an association between the Sigstad´s Score and the lowest postprandial glucose level in patients after RYGB surgery. This is investigated using a liquid mixed meal tolerance test (LMMTT). As a secondary hypothesis, associations between Edinburgh Hypoglycemia Scale (EHS) and postprandial glucose levels are investigated. Furthermore, changes of insulin and GLP-1 levels during the test are analysed. Patient characteristics including co-morbidities are studied as possible influencing parameters. Moreover, a healthy control group is included to validate the results. Finally, a flowchart/diagnostic method will be proposed for diagnosing patients who had a RYBG surgery with symptoms suggestive of PPRH. Besides the LMMTT, participants at the Ghent University Hospital will undergo additional tests such as a solid mixed meal tolerance test (SMMTT) and continuous glucose monitoring (CGM). Associations between Sigstad Score, EHS and the lowest glucose measured during CGM and SMMTT will be investigated and compared to the results of the LMMTT.

ELIGIBILITY:
Inclusion Criteria:

* for GBS group: primary GBS, 1-5 years post surgery
* for control group: 10 subjects BMI 18-25kg/m² and 10 subjects BMI >30 kg/m²

Exclusion Criteria:

* Antidiabetic medication (oral or injectable), somatostatin analogs
* Use of systemic corticosteroids
* for GBS group: Any surgery after RYGB affecting anatomic integrity of the bypass, e.g. banding, conversion of the proximal and/or distal anastomosis
* for GBS group: Any surgery before RYGB affecting anatomic integrity of the bypass, e.g. banding, conversion of the proximal and/or distal anastomosis, sleeve gastrectomy
* Known renal insufficiency: CDK ≥ 4
* Known liver cirrhosis
* Known cardiovascular risk: NYHA ≥ III
* Mental incapacity
* Language barriers with inability to communicate with research staff
* Anemia Hb < 6.2 mmol/l (10.0 g/dl)
* Cancer within < 5 years
* Pregnancy
* Allergy to the Fresubin E
* Allergy to components of the solid mixed meal (white bread, cheese spread, margarine, orange)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In total 100 GBS patients which will be recruited over multiple sites in Germany, Great Britain, Belgium and Denmark.
  Belgium will be the only site performing the solid mixed meal tolerance test and the continuous glucose monitoring additional to the liquid mixed meal tolerance test. All other sites will only do the liquid mixed meal tolerance test.
  In total 20 control patients (10 with a BMI 18-25 kg/m² and 10 with a BMI > 30 kg/m²) will be recruited. These will be recruited in Belgium (Ghent University Hospital) and the patients will undergo a liquid mixed meal tolerance test, a solid mixed meal tolerance test and a continuous glucose monitoring
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2020-05-05 (Actual); Study Completion 2020-05-05 (Actual)

PRIMARY OUTCOMES:
Association between Sigstad's score and the lowest postprandial glucose levels | end 2018
  we are investigating whether there is an association between the Sigtad's score and the lowest glucose levels postprandialy

SECONDARY OUTCOMES:
Association between Ediinburgh Hypoglycemia scale and the lowest postprandial glucose levels | end 2018
  we are investigating whether there is an association between the Ediinburgh Hypoglycemia scale and the lowest glucose levels postprandialy
flow chart for diagnosis of postprandial reactive hypoglyceamia | end 2018
  Proposing a flowchart/diagnostic method for the diagnosis of postprandial reactive hypoglycemic syndrome which occurs in people who underwent a gastric bypass surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Endocrinology, UZ Ghent Hospital, Ghent, Belgium